CLINICAL TRIAL: NCT02434315
Title: Evaluation of the FreeStyle Libre Pro for Individuals With Insulin Managed Type 2 Diabetes in Primary & Secondary Care
Brief Title: FreeStyle Libre Pro Use in Primary & Secondary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ADC-UK-PMS-14024
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Sensing Technology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A - Control (Active Comparator): FreeStyle Libre Pro 3 sensor wears
  Interventions: Device: FreeStyle Libre Pro 3 sensor wears
- Group B - Intervention (Experimental): FreeStyle Libre Pro 4 sensor wears, 2 with reviews
  Interventions: Device: FreeStyle Libre Pro 4 sensor wears, 2 with reviews
- Group C - Intervention (Experimental): FreeStyle Libre Pro 6 sensor wears, 4 with reviews
  Interventions: Device: FreeStyle Libre Pro 6 sensor wears, 4 with reviews

INTERVENTIONS:
Device: FreeStyle Libre Pro 4 sensor wears, 2 with reviews — Subjects will wear the FreeStyle Libre Pro System for 14 days. 2 period of FreeStyle Libre Pro Sensor wear for data review followed by 2 further periods of Sensor wear for time in range measurement with 28 day interval between wears.
  Arms: Group B - Intervention
Device: FreeStyle Libre Pro 6 sensor wears, 4 with reviews — Subjects will wear the FreeStyle Libre Pro System for 14 days. 4 period of FreeStyle Libre Pro Sensor wear for data review followed by 2 further periods of Sensor wear for time in range measurement with 28 day interval between wears.
  Arms: Group C - Intervention
Device: FreeStyle Libre Pro 3 sensor wears — Subjects will wear the FreeStyle Libre Pro System for 14 days. 3 periods of Sensor wear for time in range measurement over a period of approximately 8 months.
  Arms: Group A - Control

SUMMARY:
The purpose of this study is to evaluate the impact of varying amount of FreeStyle Libre Pro wear as measured by time in range.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years.
* Type 2 diabetes treated with insulin therapy for at least 6 months prior to study enrolment.
* HbA1c between 58 and 108 mmol/mol (7.5 and 12.0%) inclusive.

Exclusion Criteria:

* Age at least 18 years.
* Type 2 diabetes treated with insulin therapy for at least 6 months prior to study enrolment.
* HbA1c between 58 and 108 mmol/mol (7.5 and 12.0%) inclusive.
* Participant is currently prescribed animal insulin.
* Total daily dose of insulin (TDD) is >1.75 iu/kg at entry to the study.
* Concomitant disease or condition that may compromise patient safety including and not limited to; cystic fibrosis, severe mental illness, a diagnosed or suspected eating disorder or any uncontrolled long term medical condition.
* Has a pacemaker or any other neurostimulators.
* Currently prescribed oral, intramuscular or intravenous steroid therapy for any acute or chronic condition or requires it during the study period.
* Currently receiving dialysis treatment or planning to receive dialysis during the study.
* Women who are pregnant, plan to become pregnant or become pregnant during the study.
* Participating in another study of a glucose monitoring device or drug that could affect glucose measurements or management.
* Currently using / has previously used a sensor based Glucose Monitoring System (including retrospective glucose monitoring system) within the last 6 months.
* Currently using Continuous Subcutaneous Insulin Infusion (CSII).
* Known (or suspected) allergy to medical grade adhesives.
* In the investigator's opinion the participant is unsuitable to participate due to any other cause/reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline - time in glucose range - for penultimate sensor wear | 14 day baseline phase compared to day 172 to 187
  Within arm difference in time in range in penultimate period of sensor wear compared to baseline phase

CONTACTS AND LOCATIONS:
Locations (23):
- United Kingdom (23):
  - Atherstone Surgery, Atherstone
  - Westongrove Partnership, Aylesbury
  - Pebsham Surgery, Bexhill-on-Sea
  - Omnia Practice, Birmingham
  - Hathaway Surgery, Chippenham
  - Rowden Surgery, Chippenham
  - Pound Hill Medical Group, Crawley
  - Claremont Medical Practice, Exmouth
  - White Horse Medical Practice, Faringdon
  - Parkwood Surgery, Hemel Hempstead
  - St James Hospital,, Leeds
  - Kings College Hospital, London
  - James Cook Hospital, Middlesbrough
  - Milton Keynes Hospital, Milton Keynes
  - Greenwood and Sneinton Centre, Nottingham
  - Mortimer Surgery, Reading
  - Clifton Medical Centre, Rotherham
  - Salford Royal Hospital, Salford
  - Ashfields Primary Care Centre, Sandbach
  - The Kiltearn Medical Centre, Sandbach
  - Albany House Surgery, Wellingborough
  - Rothwell Surgery, Wellingborough
  - Friarsgate Practice, Winchester

REFERENCES:
- [Derived] Ajjan RA, Jackson N, Thomson SA. Reduction in HbA1c using professional flash glucose monitoring in insulin-treated type 2 diabetes patients managed in primary and secondary care settings: A pilot, multicentre, randomised controlled trial. Diab Vasc Dis Res. 2019 Jul;16(4):385-395. doi: 10.1177/1479164119827456. PMID 31271312